CLINICAL TRIAL: NCT04028375
Title: Clinical Study of CT and MR in Staging and Prediction of Response in Patients With Gastric Cancer
Brief Title: Study of CT and MR in the Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FSK002
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2019-07

CONDITIONS: Gastric Cancer Stage; CT; MRI; Neoadjuvant Therapy
Keywords: Gastric Cancer; MRI; MSCT; Staging; Prediction and Prognosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
It is very significant that assessing staging in gastric cancer patients before surgery, furthermore, determining the optimize surgical strategy ,predict the the efficacy of neoadjuvant therapy for patients. For patients who are ineffective in neoadjuvant therapy, surgery will be more meaningful.

It has been reported that the application of CT(computed tomography,CT) and MR(magnetic resonance,MR) in staging of gastric cancer, but not in predicting clinical response to neoadjuvant therapy for gastric cancer. Only a few studies focused on T staging using conventional MRI in gastric cancer, however , relatively new sequences in the chest deserve widely used. To develop a pre-treatment evaluation methods for TN staging in patient with gastric cancer by utilization of the new imaging methods (T2-TSE-BLADE,T2 maps, StarVIBE, iShim-DWI and high resolution CT). By analysing the relationship between TN staging and imaging features to find the imaging characteristics for TN staging, and to find the indicators of new technology and reference values for facilitate pre-treatment diagnosis of TN staging, optimize surgical strategy , predict the the efficacy of adjunctive therapy , and OS and define the range of lymph node for radiotherapy , as making personal treatment planning for gastric cancer .

DETAILED DESCRIPTION:
To explore the value of CT and MR using multiple sequences, including T2-TSE-BLADE, T2 maps StarVIBE, and iShim-DWI in evaluating the preoperative TN staging and prediction of response to neoadjuvant therapy and OS in patients with gastric cancer.

Patients with endoscopically biopsy-proven gastric cancer were prospectively enrolled for imaging on CT and a 3T MRI scanner . The MRI protocol included T2-TSE-BLADE, T2 maps,iShim-DWI(diffusion weighted imaging,DWI)and StarVIBE sequences, and so on. Patients received treatment according to NCCN guideline(the National Comprehensive Cancer Network,NCCN). Readers assigned a TN stage on CT and MRI, and post-operative pathologic confirmation was considered the gold standard.

Inter-reader agreement, the diagnostic accuracy of TN staging on CT and MRI were analyzed and compared to post-operative pathologic TN staging separately. MRI features were analyzed to find the correlation between pretreatment MRI features and response or OS. The study will include 400 patients. Inter-reader agreements of TN staging were analyzed excellent for CT and MRI. Diagnostic accuracy of CT and MRI will be calculated separately.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with preoperative pathologically con-firmed gastric cancer by endoscopy and preoperative imaging data (esophagography\CT\EUS\MRI) were included.
2. No contraindications for MRI examination. No contraindications contrast.
3. The patients participate in this study with informed consent.

Exclusion Criteria:

1. The patients couldn't performed MSCT or MR scanning or artefacts affect the evaluation.
2. The patients are extremely anxious and uncooperative about surgery or neoadjuvant therapy .
3. PatientsThe patients refuse to participate in the project.
4. Other situations considered by investigators not meet the inclusion criteria.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with endoscopically biopsy-proven gastric cancer will receive treatment
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
MSCT and MRI staging in Gastric Cancer. | up to 2 year
  To evaluate the staging of gastric cancer treated with systematic therapy through MSCT and 3 T MRI which using multiple sequences.

SECONDARY OUTCOMES:
MSCT and MRI prediction of prognosis in gastric cancer | up to 2 year
  To construct a model,a depth convolution neural network based on MSCTand multi-modal MR quantitative images which can automatically mine key images characterization, combined with imaging features and prognosis,could further help to improve the prediction of response and OS of gastric cancer treated with systematic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giganti F, Tang L, Baba H. Gastric cancer and imaging biomarkers: Part 1 - a critical review of DW-MRI and CE-MDCT findings. Eur Radiol. 2019 Apr;29(4):1743-1753. doi: 10.1007/s00330-018-5732-4. Epub 2018 Oct 2. PMID 30280246
- [Background] Pang L, Wang J, Fan Y, Xu R, Bai Y, Bai L. Correlations of TNM staging and lymph node metastasis of gastric cancer with MRI features and VEGF expression. Cancer Biomark. 2018;23(1):53-59. doi: 10.3233/CBM-181287. PMID 30010108
- [Background] Borggreve AS, Goense L, Brenkman HJF, Mook S, Meijer GJ, Wessels FJ, Verheij M, Jansen EPM, van Hillegersberg R, van Rossum PSN, Ruurda JP. Imaging strategies in the management of gastric cancer: current role and future potential of MRI. Br J Radiol. 2019 May;92(1097):20181044. doi: 10.1259/bjr.20181044. Epub 2019 Mar 5. PMID 30789792
- [Background] Zhou J, Shen J, Seifer BJ, Jiang S, Wang J, Xiong H, Xie L, Wang L, Sui X. Approaches and genetic determinants in predicting response to neoadjuvant chemotherapy in locally advanced gastric cancer. Oncotarget. 2017 May 2;8(18):30477-30494. doi: 10.18632/oncotarget.12955. PMID 27802185
- [Background] Kwee RM, Kwee TC. Role of imaging in predicting response to neoadjuvant chemotherapy in gastric cancer. World J Gastroenterol. 2014 Feb 21;20(7):1650-6. doi: 10.3748/wjg.v20.i7.1650. PMID 24587644
- [Background] Ng J, Lee P. The Role of Radiotherapy in Localized Esophageal and Gastric Cancer. Hematol Oncol Clin North Am. 2017 Jun;31(3):453-468. doi: 10.1016/j.hoc.2017.01.005. Epub 2017 Mar 22. PMID 28501087
- [Background] Al-Batran SE, Homann N, Pauligk C, Illerhaus G, Martens UM, Stoehlmacher J, Schmalenberg H, Luley KB, Prasnikar N, Egger M, Probst S, Messmann H, Moehler M, Fischbach W, Hartmann JT, Mayer F, Hoffkes HG, Koenigsmann M, Arnold D, Kraus TW, Grimm K, Berkhoff S, Post S, Jager E, Bechstein W, Ronellenfitsch U, Monig S, Hofheinz RD. Effect of Neoadjuvant Chemotherapy Followed by Surgical Resection on Survival in Patients With Limited Metastatic Gastric or Gastroesophageal Junction Cancer: The AIO-FLOT3 Trial. JAMA Oncol. 2017 Sep 1;3(9):1237-1244. doi: 10.1001/jamaoncol.2017.0515. PMID 28448662
- [Derived] Li J, Yan LL, Zhang HK, Wang Y, Xu SN, Chen XJ, Qu JR. Application of intravoxel incoherent motion diffusion-weighted imaging for preoperative knowledge of lymphovascular invasion in gastric cancer: a prospective study. Abdom Radiol (NY). 2023 Jul;48(7):2207-2218. doi: 10.1007/s00261-023-03920-2. Epub 2023 Apr 21. PMID 37085731